CLINICAL TRIAL: NCT06992531
Title: Auto-immune Contribution in Symptom-based Sensory and Autonomic Disorders
Acronym: ACSSAD
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 352817
Record Dates: First submitted 2025-05-16; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Postural Orthostatic Tachycardia Syndrome (POTS); Fibromyalgia (FM)
Keywords: Postural orthostatic Tachycardia Syndrome; Fibromyalgia Syndrome; Widespread pain; Autoantibodies; Autonomic and sensory functions
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Fibromyalgia | interventions — Surveys and Questionnaires; Restraint, Physical; Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood collection (Serum and Peripheral blood mononuclear cells) Skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PoTS with pain: Participants with PoTS with an additional diagnosis of FMS
  Interventions: Other: Questionnaire and Physical Exam; Diagnostic Test: Nerve conduction studies; Diagnostic Test: Microneurography; Diagnostic Test: Quantitative Sensory Testing; Diagnostic Test: Skin biopsy; Biological: Blood Product
- PoTS without pain: Participants with PoTS without pain
  Interventions: Other: Questionnaire and Physical Exam; Diagnostic Test: Nerve conduction studies; Diagnostic Test: Microneurography; Diagnostic Test: Quantitative Sensory Testing; Diagnostic Test: Skin biopsy; Biological: Blood Product
- FMS: Participants with FMS without dysautonomia
  Interventions: Other: Questionnaire and Physical Exam; Diagnostic Test: Nerve conduction studies; Diagnostic Test: Microneurography; Diagnostic Test: Quantitative Sensory Testing; Diagnostic Test: Skin biopsy; Biological: Blood Product
- Healthy volunteers: Healthy volunteers with no diagnosed autoimmune, chronic pain, or dysautonomia condition.
  Interventions: Other: Questionnaire and Physical Exam; Diagnostic Test: Nerve conduction studies; Diagnostic Test: Microneurography; Diagnostic Test: Quantitative Sensory Testing; Diagnostic Test: Skin biopsy; Biological: Blood Product

INTERVENTIONS:
Other: Questionnaire and Physical Exam — Standardised participant questionnaires assessing neurological symptoms, including pain (NPSI, DN4, BPI), fatigue (Fatigue Severity Scale), depression and anxiety (PHQ9 and GAD7) and autonomic dysfunction (Malmo PoTS Score and COMPASS-31).
Diagnostic Test: Nerve conduction studies — Measures how fast an electrical impulse moves through sensory and motor nerves. The test will be used to identify/rule out large fibre peripheral neuropathy.
Diagnostic Test: Microneurography — Electrophysiological technique that can record action potentials from individual peripheral nerve axons in humans. The test will be used to identify/rule out small nerve fibre dysfunction.
Diagnostic Test: Quantitative Sensory Testing — Measures psychophysical sensory perception in response to different types of stimuli, such as thermal, mechanical, pressure and vibration. The test will be used to identify/rule out nerve fibre dysfunction, by generating a quantitative sensory profile of different sensory modalities.
Diagnostic Test: Skin biopsy — Safe and minimally invasive procedure to quantify intraepidermal nerve fibres density (IENFD). Reduced IENF density is associated with small fibre neuropathy.
Biological: Blood Product — A blood sample of a maximum of 120ml will be collected from a superficial upper limb vein. Blood aliquots (50ml tubes) will then be centrifuged to separate serum from the peripheral blood cells.

SUMMARY:
Postural Orthostatic Tachycardia Syndrome (PoTS) is a condition where the heart rate increases when standing up, causing symptoms like dizziness and fainting. It primarily affects young women and can be very disabling, impacting daily life. In addition to the typical symptoms related to standing, people with PoTS also experience unexplained pain and fatigue, which worsen their quality of life. The exact causes of PoTS are still unknown, but it is often triggered by viral infections and some PoTS patients show signs of immune system involvement, such as the presence of certain autoantibodies and other autoimmune conditions. Research on other chronic pain disorders, including fibromyalgia syndrome (FMS), has found that autoantibodies can cause pain by affecting how the nerves work. This study aims to investigate if similar immune-related mechanisms are behind the widespread pain seen in PoTS. This study will also look at how PoTS affects the nervous system by testing nerve activity in participants and assessing the number of nerve fibres in the skin, to check if similar changes can be seen in mice. This study will also involve participants with fibromyalgia syndrome and healthy volunteers.

DETAILED DESCRIPTION:
Postural orthostatic tachycardia syndrome (PoTS) is characterized by increased heart rate upon standing, light-headedness, and syncope. PoTS is a highly incapacitating condition affecting more than 0.2% of the population worldwide, mostly young women. The causes of this syndrome remain unknown and are still discussed, leading to unsatisfactory diagnostic tools and a delay in the recognition of PoTS as a medical condition with clear biomarkers.

The onset of postural orthostatic tachycardia symptoms is often associated with traumatic episodes or acute viral infections. An increase in PoTS diagnostic has notably been observed in adults and children during the SARS-CoV-2 epidemic. Moreover, some characteristics present in a subset of patients, namely the presence of anti-nuclear antibodies, or ganglionic acetylcholine receptor immunoglobulins, and the high prevalence of comorbid auto-immune conditions, suggest a fundamental role of the immune system in the development of PoTS.

PoTS patients report symptoms unrelated to orthostatic intolerance, including widespread pain, muscle weakness and fatigue, which remain unexplained. These symptoms contribute to lower quality of life and impair patients' daily life.

Our group has a longstanding experience in the study of widespread pain conditions linked with autoimmunity. We have recently shown that the administration of immunoglobulins purified from fibromyalgia syndrome (FMS) and chronic regional pain syndrome (CRPS) patients replicates painful and non-painful phenotypes in mice. In contrast with the CRPS mice, where a physical injury is needed to induce hypersensitivity, intraperitoneal administration of IgG was sufficient to generate mechanical hyperalgesia and abnormal responses to non-noxious stimuli in rodents.

The passive transfer of fibromyalgia symptoms from patients to mice via IgG administration presents many advantages, amongst which is the possibility of studying immune-mediated neuronal abnormalities in isolation. Upon FMS IgG administration, we observed an accumulation of pathological IgG in dorsal root ganglia (DRG), the organs relaying sensory information perceived in peripheral organs, to the spinal cord. Interestingly, the exploration of murine DRGs cells signalling revealed an increased activity of sensory neurons, canonically responsible for mechanical and thermal sensations, but also for the perception of painful stimuli. This enhanced activity was not observed with preparation isolated from mice injected with healthy volunteer immunoglobulins.

This study has revealed immune-mediated mechanisms leading to hyperexcitability in sensory neurons and causing exacerbated pain and non-painful perception in fibromyalgia. We now intend to assess whether widespread pain, observed in PoTS patients presents a similar autoimmune pathophysiology. Moreover, we aim to investigate potential abnormalities of the autonomic system caused by the administration of PoTS IgG.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 80 years of age.
* In the capacity to understand and sign an Informed Consent Form.
* Willing and able to comply with scheduled visits and study procedures.
* Diagnostic criteria for participants:
* PoTS: following Heart Rhythm Society Expert Consensus Statement criteria, 2015, with or without comorbid FMS.
* FMS: following the American College of Rheumatology criteria 2016, with Fibromyalgia Impact Questionnaire (FIQ) exceeding 50, and with an average pain intensity exceeding 5.5.
* Healthy volunteers: no diagnosed autoimmune, chronic pain, or dysautonomia condition.

Exclusion Criteria:

* Previous diagnosis of an established autoimmune condition or dermatological conditions affecting skin afferents (e.g. psoriasis, lupus, vitiligo, dermatitis…).
* Application of local anaesthetics or steroid injections within 35 days prior to the microneurography visit.
* Current use of anticoagulant therapy.
* History of peripheral neuropathy or conditions usually associated with peripheral neuropathy, such as Diabetes Mellitus, Vitamin B12 deficiency, Lyme disease, a screen positive for hepatitis B surface antigen, hepatitis C virus antibody, or antibodies against human immunodeficiency viruses 1 and 2.
* Pregnancy.
* Difficulties in locating the nerve (i.e. nerve cannot be seen or palpated) or previously known trauma or surgery in the area innervated will be a criterion for the exclusion of the participant for this part of the study.
* History of regular alcohol consumption (exceeding 14 units per week) or recent alcohol consumption exceeding 14 units per week over the last 6 months (14 units is equivalent to 7 pints [568 mL/pint] of beer at 3.6% alcohol by volume or 6 standard glasses [176 mL/glass] of wine at 12% alcohol by volume).
* Excessive consumption of caffeinated beverages (e.g., coffee, tea, cola, energy drinks), is defined as greater than 6 servings per day (1 serving/236 mL equals approximately 120 mg of caffeine).
* A history of drug abuse or addiction within 2 years before study, current regular or recreational use of marijuana (or any cannabis derivative).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients diagnosed with PoTS (50% with comorbid FMS) 50 patients diagnosed with FMS without dysautonomia Up to 100 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Evidence of immune-mediated pain mechanisms and autonomic dysfunction | From enrollment until passive tranfer experiments are performed.
  To determine whether IgG antibodies from PoTS participants (with or without FMS) induce pain-like behaviours and autonomic abnormalities in mice, following passive transfer.

SECONDARY OUTCOMES:
Assessment of electrical activity recorded from nerve fibres in humans | From enrollment until Visit 1.
  To use microneurography to measure nerve activity in participants and identify patterns consistent with small nerve fibre dysfunction.
Evidence of small fibre neuropathy (SFN) | From enrollment until passive tranfer experiments are performed.
  To evaluate intra-epidermal nerve fibre density (IENFD) in skin biopsies from PoTS participants to identify signs of SFN; similar analysis will be conducted in mice receiving participants' IgG.
IgG binding to rodent neurons | From enrollment until passive tranfer experiments are performed.
  To test whether IgG from participants' serum binds to neurons in vitro, using cell-based assays and immunofluorescence.
Correlation between participants symptoms and IgG effects in mice | From enrollment until passive tranfer experiments are performed.
  To explore whether clinical symptom severity (e.g., pain, autonomic dysfunction) correlates with the degree of abnormality observed in mice after IgG transfer.